CLINICAL TRIAL: NCT06845150
Title: Dual-Task Training in an Immersive Environment Compared to Single Task Training in Anterior Cruciate Ligament Reconstructed Individuals
Brief Title: Combined Compared to Sequential Cognitive and Physical Training in Anterior Cruciate Ligament Reconstructed Individuals
Acronym: DUACL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient recruitment rate to reach the targeted number in June 2026
Sponsor: Michelle C. Haas (Other)
Collaborators: Kantonsspital Winterthur KSW (Other); ZHAW DIZH Fellowship Program (Unknown)
Responsible Party: Sponsor-Investigator, Michelle C. Haas, Research Associate, Zurich University of Applied Sciences
Organization: Zurich University of Applied Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: DUACL
Record Dates: First submitted 2025-02-13; First posted 2025-02-25 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Anterior Cruciate Ligament Reconstruction Rehabilitation
Keywords: motor-cognitive training; dual-task training; anterior cruciate ligament injury; return to competition
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Masking Description: concealed allocation of group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dual-task training (Experimental)
  Interventions: Other: Dual-task training
- Single task training (Active Comparator)
  Interventions: Other: Single task training

INTERVENTIONS:
Other: Dual-task training — Combined simultaneous physical and cognitive training in an immersive environment
  Arms: Dual-task training
Other: Single task training — Sequential cognitive and then physical training
  Arms: Single task training

SUMMARY:
The goal of this clinical trial is to investigate changes in cognitive and physical performance after 10 weeks of dual or single task training in anterior cruciate ligament (ACL) reconstructed individuals. The main questions it aims to answer are:

* Does cognitive performance in ACL reconstructed individuals change after multiple training sessions incorporating single versus dual-task?
* Does physical performance and intrinsic motivation for training change over the course of 10 weeks when performing single versus dual-task training sessions?
* What movement patterns do ACL reconstructed individuals show during a dual-task training in an immersive environment?

Researchers will compare a combined dual-task training (combined physical and cognitive training) to a single task training (physical and cognitive training separately) to see if there are changes on cognitive performance depending on the training type.

Participants will:

* Perform dual-task or single task training twice per week for 10 weeks
* Visit the clinic before and after the training period for tests
* Visit the movement laboratory once for analysis of movement patterns

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years old
* At least 6 months after ACL injury
* Surgically reconstructed ACL
* At least 2 hours of sports participation before the injury
* Written consent of the attending surgeon to perform intensified training methods including one-legged jumps at 6 months after surgery after the first visit
* Ability to give informed consent as documented by signature
* Ability to understand instructions in German or English
* BMI < 28 kg/m^2
* Availability to take part in at least 70% of all training sessions

Exclusion Criteria:

* Surgery on the contralateral leg during the last 12 months
* Acute or chronic musculoskeletal, neurological, or cardiopulmonary disorders
* Unadjusted vision problems
* Concussion during the last 6 months
* Pregnancy
* Breastfeeding
* Amputation
* Inflammatory pain or swelling during exercising

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2025-06-05 (Actual); Primary Completion 2025-06-12 (Actual); Study Completion 2025-10-08 (Actual)

PRIMARY OUTCOMES:
Interference | Baseline, after 5 weeks of training, after 10 weeks of training
  Measured by the difference in reaction time of congruent and incongruent stimuli of the Flanker task.
Response inhibition | Baseline, after 5 weeks of training, after 10 weeks of training
  Measured by the accuracy of Go/No-Go-stimuli

SECONDARY OUTCOMES:
Jumping performance - contact time | Baseline and after 10 weeks of training
  Contact time during jumping on force plates.
Jumping performance - peak force | Baseline and after 10 weeks of training
  Peak force during jumping on force plates.
Strength | Baseline and after 10 weeks of training
  Peak force of hamstring, quadriceps, hip abduction, and hip adduction
Intrinsic motivation | At the end of each training session (2x/week for 10 weeks)
  German version of the short scale for intrinsic motivation (Kurzskala Intrinsische Motivation). For each of the 12 items there is a 5-point Likert-Scale resulting in values of 0-4. Therefore, the total score ranges from 0 to 48. The higher the score, the higher the intrinsic motivation.
Kinematics and kinetics of the lower extremities | During dual-task training in an immersive environment
  Hip, knee, and ankle angles and moments and ground reaction forces
Kinematics and kinetics of the lower extremities | Baseline and after 10 weeks of training
  Ground reaction forces, angles and moments of hip, knee, and ankle during functional tasks

OTHER OUTCOMES:
Kujala | Baseline and after 10 weeks of training
  The German version of the 13-item Kujala questionnaire will be used for assessment of anterior knee pain. Questions involve ability to do several activities and symptoms of patients. All scores of the 13 items are summed up to give a total score ranging from 0 to 100. High scores indicate a good outcome.
ACL-Return to Sport after Injury Scale | Baseline and after 10 weeks of training
  The German version of the ACL-RSI will be used. The ACL-Return to Sport after Injury Scales includes 12 items which are each answered on a Likert-scale from 0 to 100. For the total score, individual scores of each item are added and subsequently divided by the numer of questions. Hence total score ranges from 0 to 120. High scores indicate a positive psychological evaluation.
Tegner Activity Scale | Baseline and after 10 weeks of training
  The German version of the Tegner Activity Scale including 11 different stages will be used. Each stage includes activities in sports and work of patients after ACL injury. Stages range from 0 to 10.
Socio-demographic data | Baseline
  Sex, age, time since ACL reconstruction, injury history
Subjective Cognitive Load | At the end of each training session (2x/week for 10 weeks)
  Measured by the NASA-TLX questionnaire

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - KSW Kantonsspital Winterthur, Winterthur
  - ZHAW Zurich University of Applied Sciences, Winterthur

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be shared if ethically and legally possible.